CLINICAL TRIAL: NCT06072495
Title: Etiological Study of Persistent Velopharyngeal Insufficiency in Children With Operated Velopalatine Cleft by Analysis of Velopharyngeal Motor Skills in Static and Dynamic MRI
Acronym: FENTIRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PI2021_843_0208
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Velopharyngeal Insufficiency; Real Time MRI; Cleft Palate
Keywords: Velopharyngeal Insufficiency; real time MRI; Cleft palate
MeSH Terms: conditions — Velopharyngeal Insufficiency; Cleft Palate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- child with operated isolated labial cleft (Experimental)
  Interventions: Other: real time MRI
- child with isolated operated velopalatal cleft with severe VPI ( IIB//IIM) and normal velum anatomy (Experimental)
  Interventions: Other: real time MRI
- child with isolated operated velopalatal cleft with soft VPI (I/I-II) and abnormal velum anatomy (Experimental)
  Interventions: Other: real time MRI
- child with isolated operated velopalatal cleft with normal anatomy and soft VPI (Experimental)
  Interventions: Other: real time MRI

INTERVENTIONS:
Other: real time MRI — ubjects will be scanned in the supine position using ACHIEVA 3T TX DStream Philips® and a 33 channels head and neck coil. An elastic strap will be fixed to the forehead to limits movement during scan. Headset will be used to cancel the loud MRI noise and to communicate with the subjects

SUMMARY:
Velopharyngeal insufficiency is defined as the inability of the soft palate to isolate the nasopharynx from the oropharynx. It is a frequent sequela in patients with a velopalatine cleft despite anatomical restoration of the soft palate by intravelar veloplasty at 6 months. If rehabilitation by a speech therapist is not successful, a pharyngoplasty can be discussed. In the last ten years, MRI was used in dynamic and static way, to analyzed velopharyngeal muscles, in particular Levator Veli Palatini. MRI could be used to identify the etiology of VPI in those patients, and thus allow personalized rehabilitation and surgical management. The aim of this study is to examine the differences in velopharyngeal motricity as well as velar muscles morphology, positioning, and symmetry of children with repaired cleft palate with different degrees of severity of velopharyngeal insufficiency (VPI), and children with labial cleft (noncleft palate anatomy).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 12 years with Isolated cleft lip
* isolated velopalatal cleft
* Without a diagnosis of syndromic cleft or Pierre Robin sequence
* French speaking, and French is the native language
* Operated with a cheiloplasty (for cleft lip) or an intravelar Veloplasty (according to Sommerlad) at the Amiens University Hospital
* Whose follow-up is done at the Amiens University Hospital

Exclusion Criteria:

* Refusal of the parents and/or the patient
* With a contraindication to MRI
* Whose follow-up was initiated in another center and/or whose surgery was performed in another center
* Whose surgical schedule has not been followed
* Patient with severe neurological or neuropsychiatric disorders or Severe speech and language delay not related to the cleft anatomy
* Patients treated with fixed, non-removable orthodontic treatment.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ratio between the diameter of pharynx at rest and during phonation. | day 1
closure distance between the velar knee and the posterior pharyngeal wall | day 1
distance between the velar knee and the posterior pharyngeal wall | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No